CLINICAL TRIAL: NCT05430594
Title: Long-term Followup of Children Was Born From COVID Positive Mother During Birth
Brief Title: This Study Investigate the Impact of Maternal COVID-19 Infection During Birth on the Childrens' Physical and Mental Development.
Acronym: Coronababies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Other Study IDs: SE RKEB: 14/2022.
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: followup; longterm outcome; child development; maternal COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study investigates the impact of the maternal COVID infection during birth on the children's development: physical and mental outcomes. We would like to differentiate the effect from the viral infection and effect of the pandemic period, too.

ELIGIBILITY:
Inclusion Criteria:

* postitive maternal COVID test during the birth
* the newborn was cared at the Semmelweis University after birth

Ages: 12 Months to 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Firstly we examine the infants at 1 year old. We do control examination if it is necessary or give advice. We did a next examination at 2 years old in every cases.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental outcome | 2 years old

SECONDARY OUTCOMES:
Neurodevelopmental outcome | 1 year old
Phsycosomatic outcome | 1 and 2 years old
Regulation disorders | 1 and 2 years old
Feeding | 1 and 2 years old
Maternal mental status | 1 and 2 years old

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Department of Obstetrics and Gynecology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No